CLINICAL TRIAL: NCT05833009
Title: Study on the Optimal Scheme of Acupuncture Treatment for Schizophrenia-related Central Obesity
Brief Title: Acupuncture Treatment for Schizophrenia-related Central Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Shanghai University of Traditional Chinese Medicine (Other); Yueyang Hospital of lntegrated Traditional Chinese and Western Medicine, Shanghai University of Traditional Chinese Medicine (Unknown); Shanghai Huangpu Mental Health Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-64
Record Dates: First submitted 2023-02-26; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-01

CONDITIONS: Schizophrenia; Central Obesity
MeSH Terms: conditions — Schizophrenia; Obesity, Abdominal | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Acupuncture Group (Experimental): They receive actual acupuncture on purpose acupoints.
  Interventions: Device: Acupuncture
- Sham Group (Sham Comparator): They receive actual acupuncture on points but not an acupoint around the purpose acupoints.
  Interventions: Device: Acupuncture
- non-Acupuncture Group (Sham Comparator): They receive fake acupuncture (no needle) on purpose acupoints.
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture — All the groups receive respective treatment 3 times a week for the first eight weeks, twice a week for another 8 weeks, and once a week for the last 4 weeks.

SUMMARY:
This clinical trial aims to test the effect of acupuncture in patients with schizophrenia-related central obesity. The main question it aims to answer is:

• The effect, safety, and maintenance of acupuncture on schizophrenia-related central obesity.

Participants will receive acupuncture treatment on purpose acupoints, acupuncture on acupoint peripheries, or fake acupuncture treatment on purpose acupoints for 20 weeks. And they need three follow-up visits during the treatment period and two follow-up visits after treatment.

Researchers will compare the waist circumstance of these three groups to see if the purpose acupoints are valid for schizophrenia-related central obesity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with schizophrenia (Diagnostic and Statistical Manual of Mental Disorders: Fifth Edition);
* Continuous use of antipsychotics for more than one year (may be combined with mood stabilizers, antianxiety medications, antidepressants, and benzodiazepines);
* Abdominal obesity (central obesity): waist circumference ≥90cm for men or ≥85cm for women (Chinese Standard);
* All participants and their guardians signed informed consent.

Exclusion Criteria:

* Had various traditional Chinese medicine or chemical drugs, or acupuncture treatments for central obesity within two weeks before enrollment;
* Pregnant or lactating woman;
* Organic mental disorders and mental disorders induced by psychoactive and non-addictive substances;
* With other diseases affecting their mental state (e.g., chronic obstructive pulmonary disease, coronary heart disease, angina pectoris, stroke, painful joint diseases, severe psychiatric diseases, tumors, and other physical diseases)
* Severe liver and kidney insufficiency or other serious diseases of the system;
* With a family history of metabolic diseases such as hypertension, diabetes, and hyperlipidemia;
* Acupuncture dizziness, needle phobia, and other intolerant acupuncture treatment;
* Patients who are not treated according to the regulations, cannot determine the efficacy or have incomplete data affecting the efficacy and safety evaluation.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Waist Circumference at 8 weeks, 16 weeks, 20 weeks, 32 weeks, respectively | Baseline, 8 weeks, 16 weeks, 20 weeks, 32 weeks
  Waist Circumference in centimiter

SECONDARY OUTCOMES:
Change from Baseline Body Weight Index at 8 weeks, 16 weeks, 20 weeks, 32 weeks, respectively | Baseline, 8 weeks, 16 weeks, 20 weeks, 32 weeks
  weight and height will be combined to report BMI in kg/m^2
Change from Baseline Hip Circumference at 8 weeks, 16 weeks, 20 weeks, 32 weeks, respectively | Baseline, 8 weeks, 16 weeks, 20 weeks, 32 weeks
  Hip Circumference in centimiter
Change from Baseline both Blood Pressure at 8 weeks, 16 weeks, 20 weeks, 32 weeks, respectively | Baseline, 8 weeks, 16 weeks, 20 weeks, 32 weeks
  both Blood Pressure in mm/Hg
Change from Baseline Blood Triglyceride at 16 weeks, 32 weeks, respectively | Baseline, 16 weeks, 32 weeks
  Blood Triglyceride in mmol/L
Change from Baseline Blood Total Cholesterol at 16 weeks, 32 weeks, respectively | Baseline, 16 weeks, 32 weeks
  Total Cholesterol in mmol/L
Change from Baseline Blood Low-density Lipoprotein at 16 weeks, 32 weeks, respectively | Baseline, 16 weeks, 32 weeks
  Blood Low-density Lipoprotein in mmol/L
Change from Baseline Blood High-density Lipoprotein at 16 weeks, 32 weeks, respectively | Baseline, 16 weeks, 32 weeks
  Blood High-density Lipoprotein in mmol/L
Change from Baseline Blood Glucose at 16 weeks, 32 weeks, respectively | Baseline, 16 weeks, 32 weeks
  Blood Glucose in mmol/L
Change from Baseline Positive And Negative Syndrome Scale at 8 weeks, 20 weeks, 32 weeks, respectively | Baseline, 8 weeks, 20 weeks, 32 weeks
  The Positive And Negative Syndrome Scale is used for valuation of positive symptom, negative symptom and general symptom of patients with schizophrenia. The score range of Positive And Negative Syndrome Scale is 0 to 150. The higher the score, the more severe the psychiatric symptoms.
Change from Baseline Clinical Global Impression at 8 weeks, 20 weeks, 32 weeks, respectively | Baseline, 8 weeks, 20 weeks, 32 weeks
  The Clinical Global Impression evaluates the severity of ilness, global improvement and efficacy index. The score range of severity of ilness is 0 (none) to 7 (extremly severe). The score range of global improvement is 0 (none) to 7 (seriously deteriorated). The score range of efficacy index is 0 (none) to 4 (effective and no adverse effect).
Change from Baseline Personal and Social Performance Scale at 8 weeks, 20 weeks, 32 weeks, respectively | Baseline, 8 weeks, 20 weeks, 32 weeks
  The score range of Personal and Social Performance Scale is 1 to 100. The higher score, the better personal and social performance.
Change from Baseline Appetite visual analogue scale at 8 weeks, 20 weeks, 32 weeks, respectively | Baseline, 8 weeks, 20 weeks, 32 weeks
  The score range of Appetite visual analogue scale is 0 to 10. The higher score, the better appetite.
Change from Baseline Treatment Emergent Symptom Scale at 8 weeks, 16 weeks, 20 weeks, 32 weeks, respectively | Baseline, 8 weeks, 16 weeks, 20 weeks, 32 weeks
  The Treatment Emergent Symptom Scale contains 34 different common adverse effects in psychiatry patients. Each adverse effect can be assessed from three aspects, which are serverity, relationship with medications, and mesurement taken. The score range of serverity is 0 (none) to (servere). The range of relationship with medication is none, basicly (likelihood 10%) , maybe (likelihood 10%-50%), very likely (likelihood 50%-80%), definitely (likelihood over 90%). The score range of measurement taken is 0 (none) to 5 (stop medication).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - Shanghai Huangpu Mental Health Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes